CLINICAL TRIAL: NCT02584335
Title: Randomised, Double-blind Clinical Trial to Evaluate the Reduction of Pain in the Wounds Treatment Previously Applying Lidocaine Topical Solution vs Placebo
Brief Title: To Evaluate Reduction of Pain in Wounds Treatment Previously Applying Lidocaine Topical Solution vs Placebo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with the recruitment
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Antonia Dalmau Llitjos, PhD in Anesthesiology, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013LIDO; 2013-005077-52 (EudraCT Number)
Record Dates: First submitted 2015-10-09; First posted 2015-10-22 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Wounds; Local Anesthesia
Keywords: wound treatment; lidocaine; pain reduction; local anesthetic
MeSH Terms: conditions — Wounds and Injuries | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine solution ("A") (Active Comparator): Two sterile gauzes will be dampen with the content of the second syringe (the content of the first syringe is always 20 ml of saline solution and it is the first sterile gauzes administrated always) that will contain 20ml of 0.5% lidocaine dilution when the wound treatment process is assigned to the letter "A". The nurse has a third syringe exactly like this second syringe to apply if necessary (process still painful to the patient).
  Interventions: Drug: Lidocaine solution ("A")
- Saline solution ("B") (Placebo Comparator): Two sterile gauzes will be dampen with the content of the second syringe (the content of the first syringe is always 20 ml of saline solution and it is the first sterile gauzes administrated always) that will contain 20ml of saline solution when the wound treatment process is assigned to the letter "B". The nurse has a third syringe exactly like this second syringe to apply if necessary (process still painful to the patient). In this case, the three syringes supplied to the nurse, have saline solution.
  Interventions: Drug: Saline solution ("B")

INTERVENTIONS:
Drug: Lidocaine solution ("A") — Each of 26 patients will be evaluated during 6 consecutive wound treatments. The nurse will receive 3 syringes for each procedure, the syringe 1 always contains saline solution (blinded to the patient and to the nurse) to register the basal pain; the other two syringes are identical (number 2 and 3) and contain the study drug: lidocaine solution or saline solution.
  The investigators randomise the patients depending on the administration sequence (ABABAB or BABABA). When the procedure is "A", the nurse will receive the syringes number 2 and 3 containing lidocaine solution to apply (blinded to the nurse, the patient and the doctor).
  Note: The investigators consider important apply both treatments (lidocaine solution and saline solution) alternatively to avoid the bias that could might fall a cause of wound evolution (to heal or to get worse). And it is important that the same patient receives both treatments to decrease the subjective component in pain perception.
  Arms: Lidocaine solution ("A")
Drug: Saline solution ("B") — Each of 26 patients will be evaluated during 6 consecutive wound treatments. The nurse will receive 3 syringes for each procedure, the syringe 1 always contains saline solution (blinded to the patient and to the nurse) to register the basal pain; the other two syringes are identical (number 2 and 3) and contain the study drug: lidocaine solution or saline solution.
  The investigators randomise the patients depending on the administration sequence (ABABAB or BABABA). When the procedure is "B", the nurse will receive the syringes number 2 and 3 containing saline solution to apply (blinded to the nurse, the patient and the doctor).
  Note: The investigators consider important apply both treatments (lidocaine solution and saline solution) alternatively to avoid the bias that could might fall a cause of wound evolution (to heal or to get worse). And it is important that the same patient receives both treatments to decrease the subjective component in pain perception.
  Arms: Saline solution ("B")

SUMMARY:
The purpose of this study is to evaluate if applying a lidocaine topical solution before wounds treatment decreases the pain of the procedure in comparison with placebo solution.

DETAILED DESCRIPTION:
The manipulation of the wounds for its treatment is a painful process and there is currently no marketed any topical drug to decrease this suffering.

The objective of this study is to demonstrate that lidocaine topical solution applied prior to wounds treatment, reduces the pain of the procedure compared to the treatment done after application of placebo solution. In addition, if the process was less painful, the consumption of systemic analgesics would be reduced (or eliminated) and, therefore, also its secondary effects.

It is a pilot, single-center clinical trial, prospective, randomised, double-blind, placebo-controlled study that will include 26 patients admitted in Bellvitge University Hospital (HUB) who present painful wound treatments.

The Pharmaceutical Department of HUB prepares a dilution of lidocaine 0.5% in 20ml disposable syringes and also identical disposable syringes containing 20ml saline solution (process authorized by the Spanish Agency of Medicines and Sanitary Products).

Each patient included will be subject to 6 procedures, randomised according to the sequence of treatment ABABAB or BABABA ("A" is lidocaine solution, "B" is placebo solution), according to a random list.

After a doctor of The Pain Department evaluates and includes the patient into the study, prescribes the treatment and the Pharmaceutical Department provides 3 identical syringes (numbered), for each procedure, to the nurse of the patient. The first syringe will contain always saline solution (this is unknown for the patient and the nurse) doing this, the investigators obtain the basal pain of each procedure. The other two syringes contain the studying solution (lidocaine or saline solution, according the sequence of the random list) but always the same solution in both.

The doctors of the Pain Department ask the patient about the pain before starting the procedure and determine according the "Verbal numerical scale" (VNS) from 0 to 10 points. The nurse, under sterile conditions, will dampen two sterile gauzes with the solution contained in the syringe 1, and will apply on the wound during 10 minutes before starting the treatment. After this time, the nurse starts the treatment of the wound and the doctor asks again about the pain punctuation on the VNS and register it. All this procedure is repeated with the contain of the syringe 2 and register the punctuation. If the procedure is still painful, the nurse applies (following the same procedure) gauzes with the solution contained in the syringe 3 and the doctor register the VNS punctuation. If even this third application, the treatment is still painful, each patient has prescribed a systemic analgesic to be used at this point if necessary (it does not matter which analgesic, the best for each patient, the only condition is that it can not be modified during the period of inclusion into the study, it is, 6 procedures) and the punctuation in the VNS is also registered. Furthermore, during each procedure, the nurse and the doctor, control the appearance of side effects and 7 days after the last procedure, the doctor contacts to the patient for check the clinical safety.

Comparing the procedures carried out after lidocaine solution with saline solution, the investigators will evaluate the reduction of pain in the wounds treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has accepted and signed the informed consent before the random process.
* Patients with painful wound treatments
* Wounds or sores of any aetiology (vascular insufficiency, diabetics, traumatic, postsurgical...) that implies at minimum dermis or epidermis, it is, II to IV degree in the Spanish Classification of Sores made by the "National Group to Study and Management of Pressure Ulcers and Chronic Wounds" (GNEAUPP).
* Women in fertile age with pregnancy test negative.
* Men and women in fertile age using contraceptive measures

Exclusion Criteria:

* Precedents of allergic reaction to local anesthesics type amides.
* Wounds or sores degree I on the GNEAUPP Classification (without discontinuity of skin).
* Wounds or sores too large (which require more than 40 ml of solution to cover).
* Wounds around the eyes.
* Patients who presents disturbance of cardiac conduction: atrioventricular block (second or third degree) or bifascicular block
* Patients with altered level of consciousness (Glasgow Coma Scale value less than 14)
* Patients following hemodialysis, peritoneal dialysis or continuous hemofiltration treatment.
* Patients suffering moderate or severe hepatic insufficiency.
* Pregnant or lactating women.
* Patients who refuse to participate in the study.
* Patients requiring wounds treatment more than once each day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Register the VNS punctuation during wound treatments to demonstrate pain reduction (less VNS punctuation) when lidocaine solution has been administrated comparing to placebo. | The assessment is done six times (one for each wound treatment). The time frame ranges from the date of randomization to the date than the sixth wound treatment has been done; it is up to 19 days.
  The doctor asks to the patient about the punctuation on the VNS before touching the wound and when the wound treatment starts, it is, 10 minutes later than the dampen gauzes (with the syringe 1 content) has been applied on the wound and the VNS punctuation is registered. The nurse does the same procedure with the syringe 2 content and the VNS punctuation is registered. The syringe 3 content is only applied if the procedure is still painful, and the VNS punctuation is also registered.
  This process is done during 6 consecutive wound treatments for each patient. The time frame is up to 19 days because it depends on the need of treatment of each patient: every 24, 48 or 72 hours.
  At the end of the study, the investigators, will compare the punctuation registered when lidocaine solution has been administrated with the procedures realized when placebo solution was administrated, to demonstrate if the procedure is less painful (less VNS punctuation) when lidocaine solution was applied.

SECONDARY OUTCOMES:
Register if systemic analgesics are required after the third syringe content application and compare if it decreases when lidocaine solution has been applied comparing to placebo. | The assessment is done six times (one for each wound treatment). The time frame ranges from the date of randomization to the date than the sixth wound treatment has been done; it is up to 19 days.
  If the wound treatment is still painful after application the dampen gauzes with the third syringe content, each patient has prescribed a systemic analgesic to decrease the pain. It does not matter which analgesic, the only condition is that it can not be modified during the period of inclusion into the study, it is 6 consecutive wound treatments. The time frame is up to 19 days because it depends on the need of treatment of each patient: every 24, 48 or 72 hours.
  The need of the systemic analgesic to decrease the pain, in spite of the topical solution contained in the three syringes, it is registered for each wound treatment. At the end of the study, the investigators, will assess the requirements of systemic analgesics and if it exists any relation with lidocaine solution or placebo solution.
Register the efficacy (decrease VNS punctuation) of systemic analgesics when it has been required during the wound treatment. | The assessment is done six times (one for each wound treatment). The time frame ranges from the date of randomization to the date than the sixth wound treatment has been done; it is up to 19 days.
  If the wound treatment is still painful after application the dampen gauzes with the third syringe content, each patient has prescribed a systemic analgesic to decrease the pain. It does not matter which analgesic, the only condition is that it can not be modified during the period of inclusion into the study, it is 6 consecutive wound treatments. The time frame is up to 19 days because it depends on the need of treatment of each patient: every 24, 48 or 72 hours.
  The VNS punctuation before and after systemic analgesic administration is registered. At the end of the study, the investigators will assess the efficacy (decrease VNS punctuation) of systemic analgesic comparing the VNS punctuation registered before and after the administration.
Register the requirements of systemic analgesics at 60 minutes after each procedure and compare if it decreases when lidocaine solution has been applied comparing to placebo. | The assessment is done six times (60 minutes after each wound treatment). The time frame ranges from the date of randomization to the date than the sixth wound treatment has been done; it is up to 19 days.
  At Bellvitge University Hospital, the treatment prescription and administration has an electronic registration so, the investigators have the timing of administration registered at the computer.
  The investigators will compare if the need of systemic analgesics decrease (need of administration or not need of administration) at 60 minutes after the procedure when lidocaine solution has been applied during the procedure comparing when placebo has been administrated.
Register the number of doses of rescue systemic analgesics during the next 24 hours after each procedure and compare if it decreases when lidocaine solution has been applied comparing to placebo. | The assessment is done six times (during the next 24h after each wound treatment). The time frame ranges from the date of randomization to the day after than the sixth wound treatment has been done; it is up to 20 days.
  All the patients have prescribed a fixed systemic analgesia and rescue systemic analgesia (only administrated if the patient has pain). At Bellvitge University Hospital, the treatment prescription and administration has an electronic registration so, the investigators have the drug, the dose, the route of administration (all this invariable during the patient is included into the study) and the timing registered at the computer.
  The investigators will compare if the needs (number of doses) of rescue systemic analgesics decrease during the next 24 hours when lidocaine solution has been applied during the procedure comparing when placebo has been administrated.
Register the number of applications that it is necessary to decrease the pain (less punctuation in VNS) during the wound treatment procedure (it is: 1 or 2 applications). | The assessment is done six times (one for each wound treatment). The time frame ranges from the date of randomization to the date than the sixth wound treatment has been done; it is up to 19 days.
  The content of the syringes 1 and 2 will be always applied (the number 1 contains always saline solution to register the basal pain, and the syringe 2 is the study drug: lidocaine solution or saline solution, according to the random list) and the VNS punctuation is registered after both applications. If the procedure is still painful after the content of the syringe 2 application, the content of the syringe 3 is applied (it is always the same study drug that contents the syringe 2 for each procedure) and it is registered as well as the VNS punctuation given by the patient.
  At the end of the study, the investigators will determine how many times it has been necessary to apply the third syringe to reduce the pain (less punctuation given in the VNS) and, doing this, determinate if it is necessary one or two applications of the study drug to reduce the pain.
Register if any side effects is detected. | The assessment is done six times (one for each wound treatment). The time frame ranges from the date of randomization to 7 days after the sixth wound treatment has been done; it is up to 26 days.
  Registering if any side effect (local or systemic) appears during the procedures and comparing if any relation exists with lidocaine solution.
  Seven days after the sixth procedure has been done, the investigators will contact with the patient to take care that any side effects has been detected.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Dalmau, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelone, Spain

REFERENCES:
- [Result] Ozgocmen S, Kaya A, Coskun BK. Topical lidocaine helps reduce pain of digital ulcers in systemic sclerosis (scleroderma). Clin Rheumatol. 2006 May;25(3):378-9. doi: 10.1007/s10067-005-0016-1. Epub 2005 Oct 7. No abstract available. PMID 16211339
- [Result] Franz-Montan M, Ranali J, Ramacciato JC, de Andrade ED, Volpato MC, Groppo FC. Ulceration of gingival mucosa after topical application of EMLA: report of four cases. Br Dent J. 2008 Feb 9;204(3):133-4. doi: 10.1038/bdj.2008.48. PMID 18264061
- [Result] Stahl M, Meyer C, Haas E, Glaenz T, Zutt M. Leg ulcer progression caused by topical anesthesia with EMLA cream. J Dtsch Dermatol Ges. 2008 Jul;6(7):566-8. doi: 10.1111/j.1610-0387.2007.06532.x. Epub 2007 Oct 17. English, German. PMID 17941883
- [Result] Boulinguez S, Sparsa A, Bouyssou-Gauthier ML, Bedane C, Bonnetblanc JM. Adverse effects associated with EMLA cream used as topical anesthetic for the mechanical debridement of leg ulcers. J Am Acad Dermatol. 2000 Jan;42(1 Pt 1):146-8. doi: 10.1016/s0190-9622(00)90030-6. No abstract available. PMID 10607341
- [Result] Yamashita S, Sato S, Kakiuchi Y, Miyabe M, Yamaguchi H. Lidocaine toxicity during frequent viscous lidocaine use for painful tongue ulcer. J Pain Symptom Manage. 2002 Nov;24(5):543-5. doi: 10.1016/s0885-3924(02)00498-0. PMID 12547053
- [Result] Davis MD, Adams A. Lidocaine patch for the management of leg ulcer pain. J Am Acad Dermatol. 2006 Nov;55(5 Suppl):S126-7. doi: 10.1016/j.jaad.2006.02.056. No abstract available. PMID 17052535
- [Result] Sliti N, Zaraa I, Daoud L, Trojett S, Letaief I, Mokni M, Jeddi A, Ben Osman A. [Acute bilateral palpebral necrosis: a rare complication of local anaesthesia]. Ann Dermatol Venereol. 2010 Jan;137(1):84-5. doi: 10.1016/j.annder.2009.10.001. Epub 2009 Nov 20. No abstract available. French. PMID 20110079
- [Result] Claeys A, Gaudy-Marqueste C, Pauly V, Pelletier F, Truchetet F, Boye T, Aubin F, Schmutz JL, Grob JJ, Richard MA. Management of pain associated with debridement of leg ulcers: a randomized, multicentre, pilot study comparing nitrous oxide-oxygen mixture inhalation and lidocaine-prilocaine cream. J Eur Acad Dermatol Venereol. 2011 Feb;25(2):138-44. doi: 10.1111/j.1468-3083.2010.03720.x. Epub 2010 Jun 21. PMID 20569291
- [Result] Holst RG, Kristofferson A. Lidocaine-prilocaine cream (EMLA Cream) as a topical anaesthetic for the cleansing of leg ulcers. The effect of length of application time. Eur J Dermatol. 1998 Jun;8(4):245-7. PMID 9649697
- [Result] Lok C, Paul C, Amblard P, Bessis D, Debure C, Faivre B, Guillot B, Ortonne JP, Huledal G, Kalis B. EMLA cream as a topical anesthetic for the repeated mechanical debridement of venous leg ulcers: a double-blind, placebo-controlled study. J Am Acad Dermatol. 1999 Feb;40(2 Pt 1):208-13. doi: 10.1016/s0190-9622(99)70190-8. PMID 10025747
- [Result] Bershow A, Warshaw E. Cutaneous reactions to transdermal therapeutic systems. Dermatitis. 2011 Jul-Aug;22(4):193-203. PMID 21781635
- [Result] Briggs M, Nelson EA, Martyn-St James M. Topical agents or dressings for pain in venous leg ulcers. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD001177. doi: 10.1002/14651858.CD001177.pub3. PMID 23152206
- [Result] Brolmann FE, Ubbink DT, Nelson EA, Munte K, van der Horst CM, Vermeulen H. Evidence-based decisions for local and systemic wound care. Br J Surg. 2012 Sep;99(9):1172-83. doi: 10.1002/bjs.8810. Epub 2012 Jul 6. PMID 22777856
- [Result] Cooper SM, Hofman D, Burge SM. Leg ulcers and pain: a review. Int J Low Extrem Wounds. 2003 Dec;2(4):189-97. doi: 10.1177/1534734603260556. PMID 15866847
- [Result] Sobanko JF, Miller CJ, Alster TS. Topical anesthetics for dermatologic procedures: a review. Dermatol Surg. 2012 May;38(5):709-21. doi: 10.1111/j.1524-4725.2011.02271.x. Epub 2012 Jan 13. PMID 22243434
- [Result] Descroix V, Coudert AE, Vige A, Durand JP, Toupenay S, Molla M, Pompignoli M, Missika P, Allaert FA. Efficacy of topical 1% lidocaine in the symptomatic treatment of pain associated with oral mucosal trauma or minor oral aphthous ulcer: a randomized, double-blind, placebo-controlled, parallel-group, single-dose study. J Orofac Pain. 2011 Fall;25(4):327-32. PMID 22247928
- [Result] Vanscheidt W, Sadjadi Z, Lillieborg S. EMLA anaesthetic cream for sharp leg ulcer debridement: a review of the clinical evidence for analgesic efficacy and tolerability. Eur J Dermatol. 2001 Mar-Apr;11(2):90-6. PMID 11275800